CLINICAL TRIAL: NCT02600663
Title: Identification of Patients at Risk of Chronic Back Pain Using Questionnaires
Acronym: chron_pain
Status: Terminated | Type: Observational
Why Stopped: insufficient recruitment
Sponsor: Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Other Study IDs: 2015-10
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- acute back pain

SUMMARY:
Patients with acute back pain (<6 weeks) presenting at their general practitioner will be enrolled. Patients fulfilling all inclusion criteria and showing no exclusion criteria will fill out the Heidelberg short questionnaire (HKF-R10) and the Keele STarT Back Screening Tool. These two questionnaires categorize back pain patients into individuals at risk of chronic back pain and those not at risk. Furthermore, data concerning pain location, severity, duration and impairment will be collected. Study participants will receive standard care treatment prescribed by their general practitioner. Six months later, study participants will receive a questionnaire in order to collect data concerning their present pain situation. Patients with relevant impairment in their activities of daily living as a result of back pain will be categorized as individuals with chronic back pain. Categorization at six months will be compared with the categorization at presentation.

ELIGIBILITY:
Inclusion Criteria:

* acute (<6 weeks) back pain
* >20 und <60 years of age
* good oral and written knowledge of German language

Exclusion Criteria:

* any treatment for back pain within the last 6 months
* Cauda equina
* tumor
* generalized pain
* severe systemic illness
* substance abuse
* pregnancy

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients with acute back pain presenting at the general pratcioner
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
risk of chronic back pain determined by Heidelberger short questionnaire score | at enrolment
risk of chronic back pain determined by Keele questionnaire | at enrolment

SECONDARY OUTCOMES:
numeric rating scale average pain intensity | at enrolment, at 6 months
numeric rating scale minimal pain intensity | at enrolment, at 6 months
numeric rating scale pain related sleep-loss | at enrolment, at 6 months
clothepin-algometry (numeric rating scale) | at enrolment
working days missed | at enrolment, at 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Swiss Paraplegic Centre, Nottwil, Canton of Lucerne, Switzerland

IPD SHARING:
Plan to Share IPD: No